CLINICAL TRIAL: NCT03761901
Title: REtrospective, obserVational Study to Describe the Treatment Patterns and Outcomes of Epidermal Growth Factor Receptor Mutant (EGFRm) Locally Advanced or Metastatic Non-Small-Cell Lung Cancer (NSCLC) Patients in Belgium
Brief Title: Study to Describe Treatment Patterns and Outcomes in EGFRm NSCLC Patients in Belgium
Acronym: REVEAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161R00007
Record Dates: First submitted 2018-11-16; First posted 2018-12-03 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: EGFRm; NSCLC; locally advanced; metastatic; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with EGFR mutation positive NSCLC
  Interventions: Drug: 1L treatment; Drug: 2L Treatment; Drug: 3L treatment

INTERVENTIONS:
Drug: 1L treatment — chemotherapy, EGFR TKI, immunotherapy, other
Drug: 2L Treatment — Chemotherapy, EGFR TKI, immunotherapy, other
Drug: 3L treatment — chemotherapy, EGFR TKI, immunotherapy, other

SUMMARY:
This is a retrospective, observational, multicentre study to evaluate treatment patterns and outcomes of patients diagnosed with locally advanced or metastatic EGFRm NSCLC in Belgium

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years
* Pathologically confirmed NSCLC
* Tumour harbours a mutation of EGFR
* Diagnosis (radiologically or pathologically confirmed) of locally advanced or metastatic NSCLC, not amenable to curative surgery or chemoradiotherapy between 01 September 2015 and 31 December 2017

Exclusion Criteria:

* No follow-up data available after diagnosis of locally advanced or metastatic EGFRm NSCLC
* Patients who objected to participation to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with advanced or metastatic EGFRm NSCLC between 1 september 2015 and 31 December 2017
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
demographic characteristics of patients diagnosed between 1 September 2015 and 31 December 2017 | 28 months
NSCLC characteristics at diagnosis between 1 september 2015 and 31 December 2017 | 28 months
NSCLC disease characteristics at start of 2L or 3L treatment during observation window | 36 months
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first. Descriptive statitistics will be used to analyse these endpoints.
Type of treatment received during 1L, 2L or 3L treatment during the observation window | 36 months
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first. Descriptive statitistics will be used to analyse these endpoints.
Time on treatment during 1L, 2L or 3L treatment during the observation window | 36 months
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first. Descriptive statitistics will be used to analyse these endpoints.
Proportion of patients receiving a definitive, systemic therapy for NSCLC or no definitive, systemic therapy for NSCLC/best supportive care treatment after progression on their previous therapy | 36 months
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first. Descriptive statitistics will be used to analyse these endpoints.
Reason for discontinuation after 1L, 2L or 3L treatment during observation window | 36 months
  observation window: between date of diagnosis until the data cut-off, 1 september 2018, end of clinical activity or death, whichever comes first. Descriptive statistics will be used to analyse these endpoints.
EGFR testing characteristics at diagnosis between 1 september 2015 and 31 December 2017 | 28 months
EGFR testing characteristics after progression on previous treatment | 36 months
  observation window: between date of diagnosis until the data cut-off, 01 September 2018 until end of clinical activity or death, whichever comes first. Descriptive statistics will be used to analyse these endpoints.

SECONDARY OUTCOMES:
PFS for 1L, 2L or 3L treatment during the observation window | 36 months
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first. Kaplan-Meier analysis will be used.
Time-to-treatment discontinuation for 1L, 2L and 3L treatment during the observation window | 36 months
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first. Kaplan-Meier analysis will be used.
Time to start of subsequent treatment after 1L and 2L treatment during the observation window | 36 months
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first. Kaplan-Meier analysis will be used.
OS during observation window | 36 months
  OS will be measured overall for all EGFRm NSCLC patients and depending on receipt of Osimertinib treatment and line of Osimertinib treatment.
  observation window: between date of diagnosis until the data cut-off , 01 September 2018, end of clinical activity or death, whichever comes first.
  Kaplan-Meier analysis will be used.

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (14):
  - Research Site, Antwerp
  - Research Site, Bouge
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Mechelen
  - Research Site, Mons
  - Research Site, Roeselare
  - Research Site, Sint-Niklaas
  - Research Site, Sint-Truiden
  - Research Site, Turnhout
  - Research Site, Yvoir

REFERENCES:
- [Derived] Cuppens K, Lodewyckx L, Demedts I, Decoster L, Colinet B, Deschepper K, Janssens A, Galdermans D, Pieters T; REVEAL Study Group. Real-World Treatment Patterns, Epidermal Growth Factor Receptor (EGFR) Testing and Outcomes in EGFR-Mutated Advanced Non-small Cell Lung Cancer Patients in Belgium: Results from the REVEAL Study. Drugs Real World Outcomes. 2021 Jun;8(2):141-152. doi: 10.1007/s40801-021-00243-w. Epub 2021 Mar 12. PMID 33710523
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161R00007&attachmentIdentifier=872df4e2-12ee-4617-83cd-e34e9d2877b3&fileName=REVEAL_Clinical_Study_Report_redacted_synopsis_(26_Feb_2020).pdf&versionIdentifier=